CLINICAL TRIAL: NCT00156923
Title: A Multi-Center Extension of Alkermes' Study ALK21-003-EXT (NCT01218971) to Evaluate the Long-Term Safety of Medisorb® Naltrexone
Brief Title: ALK21-010: Long-term Safety of Medisorb® Naltrexone (VIVITROL®) in Alcohol-dependent Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard L. Silverman, MD / VP, Clinical Development, Alkermes, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK21-010
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2010-12-03 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Alcoholism
Keywords: Alcohol dependence
MeSH Terms: conditions — Alcoholism | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medisorb naltrexone 380 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 380 mg
- Medisorb naltrexone 190 mg (Experimental)
  Interventions: Drug: Medisorb naltrexone 190 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 380 mg — Administered via intramuscular (IM) injection once every 4 weeks for up to 3.5 years.
  Other Names: VIVITROL® 380 mg; Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 380 mg
Drug: Medisorb naltrexone 190 mg — Administered via IM injection once every 4 weeks for up to 3.5 years.
  Other Names: Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 190 mg

SUMMARY:
This was a Phase 3, multi-center extension of Alkermes' Study ALK21-003EXT (NCT01218971) to further assess the long-term safety of repeat monthly doses of Medisorb® naltrexone (VIVITROL®).

DETAILED DESCRIPTION:
Enrolled subjects continued to receive the same dose strength of Medisorb naltrexone (ie, 190 mg or 380 mg) they had received in Study ALK21-003-EXT (NCT01218971). Assigned dose strength (high or low) was not revealed to the subject, the study investigators, or any blinded member of the clinical study team for the duration of the study period. Placebo was not administered.

ELIGIBILITY:
Primary Inclusion Criteria:

* Completed Study ALK21-003-EXT (NCT01218971), receiving all 13 injections
* Willing and able to return for scheduled clinic visits and study assessments
* Noncustodial, stable address and phone
* Written, informed consent

Primary Exclusion Criteria:

* Pregnancy or lactation
* Terminated early from study drug in Study ALK21-003-EXT (NCT01218971)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2003-10; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.

REFERENCES:
- [Result] O'Brien CP, Gastfriend DR, Forman RF, Schweizer E, Pettinati HM. Long-term opioid blockade and hedonic response: preliminary data from two open-label extension studies with extended-release naltrexone. Am J Addict. 2011 Mar-Apr;20(2):106-12. doi: 10.1111/j.1521-0391.2010.00107.x. Epub 2010 Dec 28. PMID 21314752
- See also: WHO International Clinical Trials registry platform search portal — http://apps.who.int/trialsearch/trial.aspx?trialid=NCT00156923

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who successfully completed Alkermes' Study ALK21-003EXT (NCT01218971) and who continued to meet eligibility criteria were given the option to enroll into this extension study.
Groups:
- Medisorb Naltrexone 380 mg: Administered via intramuscular (IM) injection once every 4 weeks.
- Medisorb Naltrexone 190 mg: Administered via IM injection once every 4 weeks.
Period: Overall Study
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg
Started | 56 | 52
Completed | 22 | 20
Not Completed | 34 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg | Total
Number analyzed (Participants) | 56 | 52 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 47 | 100
  >=65 years | 3 | 5 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (9.0) | 48.1 (10.0) | 46.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 37 | 32 | 69
Region of Enrollment [Number; unit: participants]
  United States | 56 | 52 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least 1 Treatment-emergent Adverse Event (TEAE)
Description: A TEAE is any adverse event (AE), whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration in this extension through the end of the follow-up period).
Time Frame: Up to 3.5 years of monthly treatment
Population: Subjects who received at least 1 injection of study drug were included in the safety analyses
Measure: Number; unit: Participants
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg
Number analyzed (Participants) | 56 | 52
Participants | 49 | 51

ADVERSE EVENTS:
Time Frame: Not including the base study (Study ALK21-003 [NCT01218958]) or the first extension (Study ALK21-003EXT [NCT01218971]), the maximum exposure to study drug and safety monitoring in subjects completing this second extension was approximately 3.5 years.
Description: AEs were summarized according to number of subjects affected as opposed to number of incidences reported for any one preferred term.
Arm/Group | Medisorb Naltrexone 380 mg | Medisorb Naltrexone 190 mg
Serious Adverse Events (participants affected / at risk) | 9/56 | 9/52
Other Adverse Events (participants affected / at risk) | 51/56 | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (N=56) | Medisorb Naltrexone 190 mg (N=52)
Alcoholism (Psychiatric disorders) | 3 | 0
Completed suicide (Psychiatric disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 1
Psychotic disorder NOS (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Coronary artery disease NOS (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Bronchitis NOS (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Meningitis viral NOS (Infections and infestations) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral arterial aneurysm (Nervous system disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Drug abuser NOS (Social circumstances) | 0 | 1
Gastric operation NOS (Surgical and medical procedures) | 1 | 0
Deep venous thrombosis NOS (Vascular disorders) | 0 | 2
Pulmonary embolism (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (N=56) | Medisorb Naltrexone 190 mg (N=52)
Upper respiratory tract infection NOS (Infections and infestations) | 13 | 11
Influenza (Infections and infestations) | 6 | 3
Nasopharyngitis (Infections and infestations) | 6 | 9
Cold symptoms (Infections and infestations) | 2 | 6
Gastroenteritis viral NOS (Infections and infestations) | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7
Rash NOS (Skin and subcutaneous tissue disorders) | 3 | 2
Toothache (Gastrointestinal disorders) | 5 | 5
Dyspepsia (Gastrointestinal disorders) | 3 | 2
Diarrhoea NOS (Gastrointestinal disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Vomiting (Gastrointestinal disorders) | 3 | 2
Alcoholism (Psychiatric disorders) | 3 | 2
Anxiety NEC (Psychiatric disorders) | 3 | 2
Insomnia (Psychiatric disorders) | 4 | 7
Depression (Psychiatric disorders) | 6 | 6
Fatigue (General disorders) | 4 | 6
Fall (General disorders) | 3 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | 4
Seasonal allergy (Immune system disorders) | 4 | 1
Headache NOS (Nervous system disorders) | 4 | 6
Dizziness (Nervous system disorders) | 3 | 2
Hypertension NOS (Vascular disorders) | 3 | 6
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days but less than or equal to 90 days from the time submitted to the sponsor for review. Revisions will be negotiated in good faith. For a multicenter study the institution/PI agree to publish/publicly present the results together with the other sites unless the sponsor grants written permission in advance.